CLINICAL TRIAL: NCT01289873
Title: Prevalence, Persistence, and Risk Factors for Oral HPV Infections in College Women
Brief Title: Prevalence, Persistence, and Risk Factors for Oral Human Papillomavirus (HPV) Infections in College Women
Acronym: HOP-IN
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Merck IISP 37942
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-08

CONDITIONS: Human Papillomavirus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine how common oral HPV infections are in college women. The investigators also will find out what risk factors are associated with having oral HPV infections. The investigators hypothesize that approximately 3% of women will have oral HPV, and that HPV will be associated with oral sexual behaviors and with smoking behaviors. Finally, for those women with oral HPV- the investigators will determine whether the infections are persistent (still present) at 3-, 6-, and 12-months after the initial diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Female
* Currently enrolled as a college student

Exclusion Criteria:

* Unable to provide an oral rinse sample
* Unable to complete survey
* Unable to provide contact information
* Already completed study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: female college students
Sampling Method: Non-Probability Sample
Enrollment: 1036 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of oral HPV | at enrollment
  any oral HPV at enrollment

SECONDARY OUTCOMES:
Persistence of oral HPV over 1 year of follow-up | 1 year
  Determine whether HPV remains present at 3-months, 6-months, and 12-months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Cook, MD, MPH, Principal Investigator — University of Florida
Locations (1):
- Student Health Care Center, Gainesville, Florida, United States